CLINICAL TRIAL: NCT05723861
Title: Virtual Reality During Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Mahdi Shamali, Postdoc Researcher, Herlev and Gentofte Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VR2023; E 19215 09 (Other: Herlev Hospital)
Record Dates: First submitted 2023-01-20; First posted 2023-02-13 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Virtual Reality; Colonoscopy
Keywords: Colonoscopy; Virtual Reality; Anxiety; Pain; Patient comfort
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR group (Experimental): Participants will receive Virtual Reality intervention in addition to routine care during colonoscopy.
  Interventions: Device: VR
- Control group (No Intervention): Receive routine treatment.

INTERVENTIONS:
Device: VR — We will use the Pico Headset, a three-dimensional Gear with a connected tablet, and will be positioned on the head with elastic straps. Patients will be instructed about the VR device before their procedure and virtual experiences will initiate just before colonoscope insertion and continuously delivered throughout the procedure for max of 20 minutes. Patients will experience max of 20 minutes of VR and if colonoscopy lasts longer than 20 min, the remaining time of colonoscopy will be performed without using VR. The visualized content of VR will be chosen by the participants among three available contents including beach, nature, or mountain with relaxing music. Participants could opt out and/or request standard medications for pain at any time before or during the procedure.
  Arms: VR group

SUMMARY:
This project will use a randomized controlled trial to test the effect of using Virtual Reality on pain, anxiety, patients' comfort, and satisfaction during colonoscopy. Patients will use a virtual reality head-mounted display and choose a visualized VR content to watch during colonoscopy. Colonoscopy will be initiated without standard sedatives and narcotics and using virtual reality distraction for as long as the patient would like (for a maximum of 20 minutes). Participants could opt out and/or request standard medications for pain at any time before or during the procedure.

DETAILED DESCRIPTION:
This project aims to investigate the clinical effectiveness and implementation potential of using VR during colonoscopy using a hybrid type 1 effectiveness-implementation design through 2 work packages. The first work package will investigate the effect of VR on pain, anxiety, patients' comfort, and satisfaction during colonoscopy using a multicenter parallel randomized controlled, open-label trial. It will also be a qualitative interview to explore the healthcare professionals' and patients' experiences with using VR during colonoscopy.

The second work package will evaluate the implementation process using mix method to understand why the intervention is (or is not) more effective than usual care, whether high intervention fidelity is achieved, what barriers and facilitators there are, how these may translate into real-world implementation, and what modifications can be made to maximize implementation success. This will be achieved using quantitative and qualitative approaches with a focus on the process evaluation around the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, and Maintenance). Quantitative (e.g., quantitative analysis of patient participation rate and reasons for refusal assessment or ineligibility) and qualitative (e.g., qualitative interview of facilitators/barriers to implementing VR) data analyses will be combined to conclude the reach, adoption, implementation, and maintenance of the intervention.

The specific aims of the project will be pursued through 2 work packages and include:

Intervention effectiveness work package Study I: To investigate the effect of VR on pain, anxiety, patients' comfort, and satisfaction during colonoscopy.

Study II: To explore the healthcare professionals' and patients' experiences with using VR during colonoscopy.

Implementation work package

Qualitative part:

1. To explore facilitators/barriers to adoption and implementing using VR during colonoscopy.
2. To explore the facilitators/barriers to sustaining using VR during colonoscopy after the study was completed.

Quantitative part:

1) To examine the potential of using VR under colonoscopy for reach and adoption.

Participants will be recruited from adult patients referred to the two outpatient Endoscopy Units. Patients who meet the inclusion criteria and give written consent will be consecutively enrolled in the trial. These patients will be randomly allocated to an experimental group (using VR), or a control group (routine care). Outcomes will be measured immediately before, after, and/or during the procedure.

Some patients in the intervention group and healthcare professionals will be asked to participate in a qualitative interview to share their experiences of using VR under colonoscopy and to evaluate the implementation process.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18
* any elective indication of colonoscopy

Exclusion Criteria:

* having visual impairments,
* having dementia
* limited Danish language skills
* a high tendency to travel sickness
* having skin disease in the facial area
* having epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Patient pain before colonoscopy procedure | 5 - 15 minutes before starting colonoscopy.
  Patients will rate their pain using an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (highest imaginable pain).
Patient pain during colonoscopy procedure | During the colonoscopy procedure (from the time colonoscopy is started until ended).
  Patients will rate their pain using an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (highest imaginable pain).
Patient pain after colonoscopy procedure | 5 - 15 minutes after the colonoscopy is ended.
  Patients will rate their pain using an 11-point numeric rating scale (NRS) ranging from 0 (no pain) to 10 (highest imaginable pain).
Patient anxiety before colonoscopy procedure | 5 - 15 minutes before starting colonoscopy.
  Patient anxiety will be measured by the short form of the State Trait Anxiety Inventory (STAI) which has five items with a 4-point Likert-type scale ranging from 0 to 3.
Patient anxiety after colonoscopy procedure | 5 - 15 minutes after the colonoscopy is ended.
  Patient anxiety will be measured by the short form of the State Trait Anxiety Inventory (STAI) which has five items with a 4-point Likert-type scale ranging from 0 to 3.
Patient comfort during colonoscopy procedure | During the colonoscopy procedure (from the time colonoscopy is started until ended).
  Patient comfort will be measured by a nurse/researcher using the five-point Modified. Gloucester Comfort Scale (MGCS) ranging from 1 (no discomfort) to 5 (severe discomfort).
Patient comfort after colonoscopy procedure | 5 - 15 minutes after the colonoscopy is ended.
  Patient comfort will be measured by a nurse/researcher using the five-point Modified. Gloucester Comfort Scale (MGCS) ranging from 1 (no discomfort) to 5 (severe discomfort).

SECONDARY OUTCOMES:
Patient satisfaction | 5 - 15 minutes after the colonoscopy is ended.
  Patient satisfaction with the procedure will be measured using an 11-point numeric rating scale ranging from 0 (no satisfaction at all) to 10 (definitely satisfied).
Patient / healthcare professional experience with using VR during colonoscopy | 30 minutes - one week after the procedure
  Qualitative interview of some patients in the intervention group and and healthcare professionals.

CONTACTS AND LOCATIONS:
Overall Officials: Mahdi Shamali, PhD, Principal Investigator — Herlev and Gentofte University Hospital; Hanne Konradsen, PhD, Principal Investigator — Herlev and Gentofte University Hospital
Locations (1):
- Department of Gastroenterology, Herlev and Gentofte Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shamali M, Vilmann P, Johansen NR, Konradsen H. Virtual reality intervention to improve quality of care during colonoscopy: a hybrid type 1 randomized controlled trial. Gastrointest Endosc. 2024 Nov;100(5):914-922.e2. doi: 10.1016/j.gie.2024.05.023. Epub 2024 Jun 6. PMID 38851457